CLINICAL TRIAL: NCT05521529
Title: Effects of CORtisol Excess and REmission in Cushing's Syndrome Over Time (CORRECT): A Prospective Non-interventional Cohort Study
Brief Title: Cushing's Syndrome Before and After Treatment (CORRECT)
Acronym: CORRECT
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-41-22
Record Dates: First submitted 2022-08-16; First posted 2022-08-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Cushing Syndrome
Keywords: Circadian Rhythm; Quality of Life
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Whole blood drawn into K-EDTA tubes and stored at -80 degrees celsius
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: no intervention, as this is an observational study — no intervention

SUMMARY:
The purpose of this study is to prospectively study patients with Cushing's syndrome before and after treatment, with a special emphasis on physical function, quality of life, and circadian rhythms.

The hypotheses are:

* Cushing's syndrome negatively impacts health-related quality of life (HRQoL) and physical functioning
* Cushing's syndrome is associated with altered circadian rhythms at the whole body level and in peripheral target tissues.
* These complications partially reverse following disease control.

ELIGIBILITY:
Inclusion Criteria:

* New (≤ 2 months) diagnosis of Cushing's syndrome (CS) of endogenous etiology:

  * ACTH-dependent CS
  * ACTH-independent CS
* Age >18 years
* Written informed consent

Exclusion Criteria:

* Active cancer
* Iatrogenic or malignant cause of CS such as adrenocortical carcinoma
* Chronic heart failure (New York Heart Association class IV)
* Chronic kidney disease Chronic Kidney Disease stage ≥3 (eGFR >30 ml/min)
* Liver disease in the form of cirrhosis
* Deemed unable to complete the study safely by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed Cushing's Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Change in CushingQoL-score | Baseline, 3 months after and 1 year after treatment
  Questionnaire filled out by patients

SECONDARY OUTCOMES:
Change in blood pressure | Baseline, 3 months after and 1 year
  Blood pressure, both standard office readings and as AOBP (Automated Office Blood Pressure)
Change in arterial stiffness and endothelial function. | Baseline, 3 months after and 1 year
  Arterial stiffness is assessed as Carotid-femoral PWV (cfPWV), measured using the SphygmoCor device (version 9; AtCor Medical
Change in endothelial function. | Baseline, 3 months after and 1 year
  Endothelial function will be assessed by the EndoPAT® device (Itamar Medical)
Change in Insulin resistance | Baseline, 3 months after and 1 year
  Assessed through fasting blood levels of insulin and glucose (Homeostasis Model Assessment, HOMA)
Change in Hba1C | Baseline, 3 months after and 1 year
  Assessed as glycated hemoglobin A1C levels measured at three time points
Change in Messenger RNA expression of core clock genes in blood leukocytes and biopsies of skeletal muscle and adipose tissue. | Baseline, 3 months after and 1 year
  Messenger RNA expression of core clock genes such as BMAL1, CLOCK, PER1-3, CRY1-2, REV-ERBα -β and -γ, RORA-C will be determined. For comparison, housekeeping genes such as Glyceraldehyde-3-phosphate dehydrogenase (GAPDH), β2 microglobulin (B2M) and β-actin (ACTB) will be used.
  All will be expressed as -fold change from baseline expression levels
Change in body composition | Baseline, 3 months after and 1 year
  Dual X-ray absorptiometry (DXA), is used to measure whole body lean body mass, and fat mass in gram
Change in Bone Mineral Density | Baseline, 3 months after and 1 year
  Dual X-ray absorptiometry (DXA), bone mineral density (BMD) of the lumbar spine and femoral neck.
Change in Vertebral Fracture Assessment | Baseline, 3 months after and 1 year
  Dual X-ray absorptiometry (DXA), is used to assess vertebral fractures (VFA).
Change in weight | Baseline, 3 months after and 1 year
  Change in weight in kilograms
Change in BMI | Baseline, 3 months after and 1 year
  Height and weight are combined to express body mass index (BMI, kg/m2)
Change in waist circumference | Baseline, 3 months after and 1 year
  waist circumference is recorded with measuring tape.
Change in hip circumference | Baseline, 3 months after and 1 year
  Hip circumference is recorded with measuring tape.
Change in Timed up and go (TUG)-test | Baseline, 3 months after and 1 year
  The TUG Test combines measures of physical performance and coordination. The TUG test measures the time to stand up, walk 3 m in a straight line, and immediately return to the chair.
  The result is expressed as the fastest time in seconds
Change in Short Physical Performance Battery (SPPB) and chair rising test - score | Baseline, 3 months after and 1 year
  The short physical performance battery (SPPB) is a group of bed-side measures that combines the results of walking speed, chair stand and balance tests.
  The result is expressed as a collective score from 0-12
Change in Handgrip strength | Baseline, 3 months after and 1 year
  Handgrip strength is measured using a hand dynamometer with the participant seated
Change in total physical activity | Baseline, 3 months after and 1 year
  Measured with an Actigraph tri-axial accelerometer on the non-dominant wrist. Expressed as Counts/day
Change in Sedentary time | Baseline, 3 months after and 1 year
  Measured with an Actigraph tri-axial accelerometer on the non-dominant wrist. Expressed as hours/day
Change in total sleep time | Baseline, 3 months after and 1 year
  Measured with an Actigraph tri-axial accelerometer on the non-dominant wrist. Expressed as hours/day
Change in IPAQ-S7S | Baseline, 3 months after and 1 year
  The questionnaire records types and intensity of physical activity and consists of seven open items
FACS of blood leukocytes | Baseline, 3 months after and 1 year
  Flow assisted cell sorting (FACS) will be performed on blood leukocytes followed by real time quantitative polymerase chain reaction on distinct cells or in single cell suspension from relevant tissue.
Change in 24 hour urinary free cortisol | Baseline, 3 months after and 1 year
  free cortisol
Change in 24 hour urinary steroid metabolome | Baseline, 3 months after and 1 year
  Steroid metabolome
Change in 24 hour urinary adreneric metabolites | Baseline, 3 months after and 1 year
  Adrenergic metabolites
Change in Hospital Anxiety and Depression Scale (HADS) score | Baseline, 3 months after and 1 year after treatment
  Questionnaire filled out by patients
Change in Single item Sleep Quality Scale (SQS) score | Baseline, 3 months after and 1 year
  Questionnaire filled out by patients

OTHER OUTCOMES:
Change in coagulation and inflammation markers in blood | Baseline, 3 months after and 1 year
  Such as ADAM17 (Tumor necrosis factor-α-converting enzyme - TACE) Soluble CD16 (Human Low affinity immunoglobulin gamma Fc region receptor III-A) Fibrinogen vWF D-dimer Plasminogen, plasminogen activator inhibitor 1 Plasmin inhibitor
Change in metabolic and cardiovascular markers in blood | Baseline, 3 months after and 1 year
  Such as plasma levels of Adiponectin, Leptin, Free fatty acids, cholesterol
Change in cytokines levels in blood | Baseline, 3 months after and 1 year
  Such as Interleukin 6 Interleukin 10 Tumor necrosis factor alfa Transforming growth factor alfa
  Measured with cytokine luminex
Participant records: Number of infections, prescriptions for antibiotics | Baseline, 3 months after and 1 year
  Assessed via electronic patient records

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto Lunde Jørgensen, Professor, Study Director — AARHUS UNIVERSITY HOSPITAL, Medical Research Laboratory
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus, State, Denmark

IPD SHARING:
Plan to Share IPD: No